CLINICAL TRIAL: NCT00314938
Title: A Double Blind, Single Dose Study To Explore The Safety, Pharmacokinetics And Pharmacodynamics Of PHA-794428 In Pediatric Patients With Growth Hormone Deficiency
Brief Title: A Single Dose Study to Evaluate the PK-PD Response and Safety of PHA-794428 in Children With Growth Hormone Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6391004
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PHA-794428

SUMMARY:
This will be the first clinical study of the development of PHA-794428 in a pediatric population. Since differences in PK and/or PD response may occur between adult and pediatric subjects, it is deemed appropriate to first conduct an exploratory single dose study in pediatric patients to assess safety and tolerability in this patient population. In addition this will add pediatric data to facilitate the prediction of the optimal therapeutic dose to be tested in repeated dose phase 2b trials in children, using PK/PD modeling

DETAILED DESCRIPTION:
The study terminated on 10-Dec-2007. Pfizer's decision to terminate the program was due to cases of injection-site lipoatrophy that were reported in the clinical Phase 2 studies after a single injection of PHA 794428.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male and female children with a minimum age of 6 years
* 2. Prepubertal as defined by Tanner staging
* 3. Growth hormone deficiency

Exclusion Criteria:

* 1. PGHD patients with uncontrolled pituitary tumor growth
* 2. Tumors within 3 mm of the optic chiasm
* 3. Serum ALT and/or AST >= 1.5 times the upper limit of normal range

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
PK, IGF-1 and safety measurements up to 2 weeks after dosing

SECONDARY OUTCOMES:
Antibody and IGFBP-3 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
- Pfizer Investigational Site, Paris, France
- Pfizer Investigational Site, Erlangen, Germany
- Pfizer Investigational Site, Petah Tikva, Israel, Israel
- Pfizer Investigational Site, Cardiff, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6391004&StudyName=A%20single%20dose%20study%20to%20evaluate%20the%20PK-PD%20response%20and%20safety%20of%20PHA-794428%20in%20children%20with%20growth%20hormone%20deficiency